CLINICAL TRIAL: NCT02858609
Title: Improving the Diagnosis of Diarrhoea in Emergency Rooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-44
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2022-10

CONDITIONS: Diarrhoea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Diarrhoea (Experimental): Patients admitted in emergency room with Diarrhoea
  Interventions: Other: Nasopharyngeal Swab

INTERVENTIONS:
Other: Nasopharyngeal Swab

SUMMARY:
A point-of-care laboratory (POC) was set at North Hospital, Marseille, France for the diagnosis in less than two hours of diarrhoea caused by known pathogens, close to the reception of Emergency service. In this instance 30% of patients have no etiological diagnosis after the POC diarrhoea tests . This lab has discovered over 200 new species of bacteria in humans, including vector bacteria and opened the field of large Deoxyribonucleic Acid (DNA ) viruses. Also, the laboratory of emerging viruses discovered many Ribonucleic Acid (RNA) viruses transmitted by arthropods. Based on this collection of new pathogens described in POC laboratory, this study proposes to expand the etiological diagnosis strategy of diarrhoea after POC tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted at hospital for diarrhoea requiring, for the emergency physician, a microbiological examination with a "POC diarrhoea kit."
* Patient who has freely signed the informed written consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Pregnant woman, parturient or nursing
* Adult major under guardianship
* Patient deprived of liberty under court order
* Patient refusing or unable to sign the informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients admitted in emergency rooms for diarrhoea with confirmed etiological diagnosis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided